CLINICAL TRIAL: NCT05249153
Title: The Effect of Combination of Dexmedetomidine and Sufentanil in Patient-controlled Intravenous Analgesia on Pediatric Patients Undergoing Scoliosis Surgery
Brief Title: Dexmedetomidine and Sufentanil Effect in PCA on Pediatric Patients Undergoing Scoliosis Surgery
Acronym: DEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZS-2546
Record Dates: First submitted 2022-01-21; First posted 2022-02-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-02

CONDITIONS: Dexmedetomidine
Keywords: dexmedetomidine; pediatric anesthesia; patient-control analgesia; scoliosis orthopedics
MeSH Terms: interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sufen (No Intervention): PCIA: continue with 0.05ug/kg/h sufentanil, 0.05ug/kg sufentainil bolus
- Sufen with low DEX (Experimental): PCIA: continue with 0.05ug/kg/h sufentanil and 0.05ug/kg/h dexmedetomidine, 0.05ug/kg/h sufentanil and 0.05ug/kg/h dexmedetomidine bolus
  Interventions: Drug: low dose of dexmedetomidine with sufentanil
- Sufen with high DEX (Experimental): PCIA: continue with 0.05ug/kg/h sufentanil and 0.1ug/kg/h dexmedetomidine, 0.05ug/kg/h sufentanil and 0.1ug/kg/h dexmedetomidine bolus
  Interventions: Drug: high dose of dexmedetomidine with sufentanil

INTERVENTIONS:
Drug: low dose of dexmedetomidine with sufentanil — low dose of dexmedetomidine in PCIA (0.05ug/kg/h sufentanil with 0.05ug/kg/h dexmedetomidine infusion, 0.05ug/kg sufentanil with 0.05ug/kg dexmedetomidine bolus)
  Other Names: Sufen with low DEX
  Arms: Sufen with low DEX
Drug: high dose of dexmedetomidine with sufentanil — high dose of dexmedetomidine in PCIA (0.05ug/kg/h sufentanil with 0.1ug/kg/h dexmedetomidine infusion, 0.05ug/kg sufentanil with 0.1ug/kg dexmedetomidine bolus)
  Other Names: Sufen with high DEX
  Arms: Sufen with high DEX

SUMMARY:
The primary purpose of this three-arm single center, randomized, subject and assessor blind, controlled clinical study is to evaluate the effect of dexmedetomidine on patient-controlled intravenous analgesia after pediatric scoliosis orthopedics.

DETAILED DESCRIPTION:
The study is a single center, randomized, subject and assessor blinded, controlled clinical study.

Children who meet the inclusion/exclusion criteria will be evaluated. The patients will use a postoperative analgesic pump which is named as patient-control-analgesia (PCA) until the end of surgery with different dose of drugs. The control group will be set as using sufentanil only (0.05ug/kg/h infusion and 0.05ug/kg bolus). The experimental group will use sufentanil combined with different doses of dexmedetomidine. Low dose of dexmedetomidine PCA formula is 0.05ug/kg/h sufentanil with 0.05ug/kg/h dexmedetomidine infusion and 0.05ug/kg sufentanil with 0.05ug/kg dexmedetomidine bolus. High dose of dexmedetomidine PCA formula is 0.05ug/kg/h sufentanil with 0.1ug/kg/h dexmedetomidine infusion and 0.05ug/kg sufentanil with 0.1ug/kg dexmedetomidine bolus.

Then patients will be followed until they discharge.

The purpose of this trial is to evaluate the effect of of dexmedetomidine on patient-controlled intravenous analgesia after pediatric scoliosis orthopedics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 1-14 years scheduled to receive scoliosis orthopedics under general anesthesia;
* Weight is ±15% of standard weight (standard weight (kg) = height (cm) -100);
* Informed consent signed.

Exclusion Criteria:

* Allergy to dexmedetomidine;
* Obvious abnormalities of heart, lung, liver, renal function and endocrine function;
* Patients who can not cooperate with this trial.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2020-09-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative opioid analgesic dosage | 48 hours postoperatively
  the total opioid consumption in PCIA postoperatively

SECONDARY OUTCOMES:
Intraoperative opioid analgesic dosage | Intraoperative
  Intraoperative opioid analgesic dosage
Effective pressing times of PCIA | 48 hours postoperatively
  extract the data from the electric analgesic pump
Total pressing times of PCIA | 48 hours postoperatively
  extract the data from the electric analgesic pump
Remedial analgesics dosage | 48 hours postoperatively
  extract the data from the followup
postoperative pain | 48 hours postoperatively
  using VAS method to evaluate pain status. 0 score refers to comfort, 10 score refers to excruciating pain. Higher scores mean a worse outcome.
LOS | through study completion, an average of 7 days postoperatively.
  the length of stay
Patient satisfaction | 48 hours postoperatively
  patients' and relatives' satisfaction, 0 score refers to dissatisfaction, 10 score refers to satisfaction. Higher scores mean a better outcome.
Nausea | 4 hours postoperatively
  Using VRS (Verbal Rating Scales) to evaluate the degree of nausea. 0 score refers to comfort, 10 score refers to excruciating nause. Higher scores mean a worse outcome.
Nausea | 8 hours postoperatively
  Using VRS (Verbal Rating Scales) to evaluate the degree of nausea. 0 score refers to comfort, 10 score refers to excruciating nause. Higher scores mean a worse outcome.
Nausea | 24 hours postoperatively
  Using VRS (Verbal Rating Scales) to evaluate the degree of nausea. 0 score refers to comfort, 10 score refers to excruciating nause. Higher scores mean a worse outcome.
Nausea | 48 hours postoperatively
  Using VRS (Verbal Rating Scales) to evaluate the degree of nausea. 0 score refers to comfort, 10 score refers to excruciating nause. Higher scores mean a worse outcome.
Nausea | 72 hours postoperatively
  Using VRS (Verbal Rating Scales) to evaluate the degree of nausea. 0 score refers to comfort, 10 score refers to excruciating nause. Higher scores mean a worse outcome.
Sedation | 4 hours postoperatively
  Using RSAS(Riker Sedation Agitation Scale) to evaluate the status of sedation. 1 score is not aroused, 2 score is very calm, 3 score is calm, 4 score is quiet cooperation, 5 is mildly agitated, 6 score was moderate agitation, and 7 score was severe agitation. Higher and lower scores both mean a worse outcome.
Sedation | 8 hours postoperatively
  Using RSAS(Riker Sedation Agitation Scale) to evaluate the status of sedation. 1 score is not aroused, 2 score is very calm, 3 score is calm, 4 score is quiet cooperation, 5 is mildly agitated, 6 score was moderate agitation, and 7 score was severe agitation. Higher and lower scores both mean a worse outcome.
Sedation | 24 hours postoperatively
  Using RSAS(Riker Sedation Agitation Scale) to evaluate the status of sedation. 1 score is not aroused, 2 score is very calm, 3 score is calm, 4 score is quiet cooperation, 5 is mildly agitated, 6 score was moderate agitation, and 7 score was severe agitation. Higher and lower scores both mean a worse outcome.
Sedation | 48 hours postoperatively
  Using RSAS(Riker Sedation Agitation Scale) to evaluate the status of sedation. 1 score is not aroused, 2 score is very calm, 3 score is calm, 4 score is quiet cooperation, 5 is mildly agitated, 6 score was moderate agitation, and 7 score was severe agitation. Higher and lower scores both mean a worse outcome.
Sedation | 72 hours postoperatively
  Using RSAS(Riker Sedation Agitation Scale) to evaluate the status of sedation. 1 score is not aroused, 2 score is very calm, 3 score is calm, 4 score is quiet cooperation, 5 is mildly agitated, 6 score was moderate agitation, and 7 score was severe agitation. Higher and lower scores both mean a worse outcome.
Vomiting | 4 hours postoperatively
  the times of vomiting
Vomiting | 8 hours postoperatively
  the times of vomiting
Vomiting | 24 hours postoperatively
  the times of vomiting
Vomiting | 48 hours postoperatively
  the times of vomiting
Vomiting | 72 hours postoperatively
  the times of vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Yuguang Huang, MD, Study Chair — Anesthesiology of PUMCH
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No